CLINICAL TRIAL: NCT02512575
Title: A Phase I, Randomized, Single-Blind, Placebo-Controlled Study To Assess The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Single Ascending Oral Doses Of AZD9567 In Healthy Subjects.
Brief Title: A Single Ascending Dose Study To Assess The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of AZD9567.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D6470C00001; 2015-002002-37 (EudraCT Number)
Record Dates: First submitted 2015-07-06; First posted 2015-07-31 (Estimated); Results first posted 2018-10-04 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-09

CONDITIONS: Safety; Tolerability; Pharmacokinetics; Pharmacodynamics; Healthy Subjects; Rheumatoid Arthritis
Keywords: AZD9567; Healthy subjects; Phase 1; placebo controlled; single ascending dose; Pharmacokinetics; Pharmacodynamics; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- AZD9567 oral suspension (Experimental): In Part A: up to 8 cohorts with single ascending doses (starting at 2 mg up to 155 mg).
  In Part B: one cohort with a single dose
  Interventions: Drug: AZD9567 Monohydrat
- Placebo (Placebo Comparator): Subjects randomized to placebo in the first 8 cohorts will receive the same dose volume of oral suspension as subjects on AZD9567 and subjects randomized to placebo in cohort 9(prednisolone cohort) will receive the same number of capsules as subjects on prednisolone.
  Interventions: Drug: Placebo oral suspension/ Placebo capsule
- Prednisolone capsules (Experimental): Within each cohort 6 subjects will be randomized to receive prednisolone 60mg oral capsules and 2 subjects randomized to receive matching placebo in a fasted state.
  Sentinel dosing will not be employed for the prednisolone cohort. The SRC will not be required to evaluate the prednisolone cohort. This cohort can be performed at any time during clinical execution of the study provided the protocol amendment was approved.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: AZD9567 Monohydrat — AZD9567 oral suspension 0.5 to 10 mg/ml
  Arms: AZD9567 oral suspension
Drug: Placebo oral suspension/ Placebo capsule — Matching placebo
  Arms: Placebo
Drug: Prednisolone — Prednisolone 60mg oral capsules (12 capsules of 5 mg each).
  Arms: Prednisolone capsules

SUMMARY:
This is a Phase I, first-in-human (FIH), randomized, single-blind, placebo-controlled, single ascending dose sequential group study in healthy male subjects. The objectives are to study the safety, tolerability, pharmacokinetics and effects on glucose homeostasis (pharmacodynamics) of AZD9567, an oral differentiated non-steroidal selective glucocorticoid receptor modulator (SGRM). The study will also assess the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of prednisolone 60 mg in comparison with high doses of AZD9567 and placebo.

DETAILED DESCRIPTION:
This is a Phase I, first-in-human (FIH), randomized, single-blind, placebo-controlled, single ascending dose sequential group study in healthy male subjects. The objectives are to study the safety, tolerability, pharmacokinetics and effects on glucose homeostasis (pharmacodynamics) of AZD9567. Additional exploratory variables (Inflammation biomarkers, ECG modelling and taste assessment) will also be evaluated. The study will also assess the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of prednisolone 60 mg in comparison with high doses of AZD9567 and placebo. The study will be conducted at a single study centre with a planned number of subjects of up to 72 healthy males, aged 18 to 55 years.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy male subjects aged 18 to 55 years with suitable veins for cannulation or repeated venipuncture.
* Have a body mass index (BMI) between 18 and 29.9 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
* Normal OGTT at screening (<7.8 mmol/L).
* Serum cortisol levels within normal limits at screening (collected as part of the clinical chemistry panel).
* Able to understand, read and speak the German language.

Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* History or presence of gastrointestinal (GI), hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* History of or active or latent tuberculosis (TB), or at risk for having acquired TB (social workers or prison staff in countries with endemic rates of TB, having lived with patients with known TB).
* History suggesting abnormal immune function, as judged by the investigator.
* Any contraindications to be treated with prednisolone (allergy to any ingredient, systemic fungal infection, certain type of malaria, inflammation of the optic nerve, or herpes infection of the eye, scheduled to have a live or attenuated live vaccination or taking mifepristone).
* History of severe affective disorder including depressive or manic-depressive illness them self or first degree relatives.
* History of previous steroid psychosis
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
* Any latent or chronic infections (e.g., recurrent sinusitis, genital or ocular herpes, urinary tract infection) or at risk of infection (surgery, trauma, or significant infection), or history of skin abscesses within 90 days prior to the first administration of IMP.
* Any clinically important laboratory abnormalities (clinical chemistry, hematology, coagulation or urinalysis results), as judged by the investigator. In particular a subject with an abnormal value in alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transpeptidase (GGT), creatinine, thyroid-stimulating hormone (TSH), fasting glucose, International Normalised Ratio (INR), haemoglobin (Hb), white blood cell (WBC), absolute neutrophil or platelet count will be excluded.
* Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV).
* Abnormal vital signs, after 10 minutes supine rest, defined as any of the following: Systolic BP (SBP) < 90mmHg or ≥ 140 mmHg, Diastolic BP (DBP) < 50mmHg or ≥ 90 mmHg, Pulse < 45 or > 85 beats per minute (bpm).
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting ECG and any clinically important abnormalities in the 12-lead ECG, as considered by the investigator that may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology, particularly in the protocol defined primary lead or left ventricular hypertrophy.
* Prolonged QTcF > 450 ms or family history of long QT syndrome.
* PR(PQ) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation).
* PR (PQ) interval prolongation (> 240 ms) intermittent second (Wenckebach block while asleep is not exclusive) or third degree AV block, or AV dissociation

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2016-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainhard Fuhr, Dr. med., Principal Investigator — PAREXEL International GmbH, Berlin
Locations (1):
- Research Site, Berlin, Germany

REFERENCES:
- [Derived] Hegelund Myrback T, Prothon S, Edman K, Leander J, Hashemi M, Dearman M, Edenro G, Svanberg P, Andersson EM, Almquist J, Ammala C, Hendrickx R, Taib Z, Johansson KA, Berggren AR, Keen CM, Eriksson UG, Fuhr R, Carlsson BCL. Effects of a selective glucocorticoid receptor modulator (AZD9567) versus prednisolone in healthy volunteers: two phase 1, single-blind, randomised controlled trials. Lancet Rheumatol. 2020 Jan;2(1):e31-e41. doi: 10.1016/S2665-9913(19)30103-1. Epub 2019 Dec 9. PMID 38258274

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 1, single-center (Berlin), randomized, single-blind, placebo-controlled study carried on 72 healthy male participants (8 subjects per cohort). In Cohort 1-8, participants were randomized to AZD9567:placebo (6:2). In Cohort 9, participants were randomized to prednisolone:placebo (6:2). Participants received treatment in a fasted state
Pre-assignment Details: Screening period (Day -28 to Day -3). For Cohort 7, screening period was up to 21 days
Groups:
- AZD9567 - 2 mg: In Cohort 1, participants received single dose of AZD8567 2 mg oral suspension in the fasted state
- AZD9567 - 10 mg: In Cohort 2, participants received single dose of AZD8567 10 mg oral suspension in the fasted state
- AZD9567 - 20 mg: In Cohort 3, participants received single dose of AZD8567 20 mg oral suspension in the fasted state
- AZD9567 - 40 mg: In Cohort 4, participants received single dose of AZD8567 40 mg oral suspension in the fasted state
- AZD9567 - 80 mg: In Cohort 5, participants received single dose of AZD8567 80 mg oral suspension in the fasted state
- AZD9567 - 100 mg: In Cohort 6, participants received single dose of AZD8567 100 mg oral suspension in the fasted state
- AZD9567 - 125 mg: In Cohort 7, participants received single dose of AZD8567 125 mg oral suspension in the fasted state
- AZD9567 - 155 mg: In Cohort 8, participants received single dose of AZD8567 155 mg oral suspension in the fasted state
- Prednisolone - 60 mg: In Cohort 9, participants received orally single dose of prednisolone 60 mg capsule in the fasted state
- Pooled Placebo: In Cohort 1-8, participants were randomized to AZD9567:placebo (6:2). In Cohort 9, participants were randomized to prednisolone:placebo (6:2)
Period: Overall Study
Arm/Group | AZD9567 - 2 mg | AZD9567 - 10 mg | AZD9567 - 20 mg | AZD9567 - 40 mg | AZD9567 - 80 mg | AZD9567 - 100 mg | AZD9567 - 125 mg | AZD9567 - 155 mg | Prednisolone - 60 mg | Pooled Placebo
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 18
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 18
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD9567 - 2 mg | AZD9567 - 10 mg | AZD9567 - 20 mg | AZD9567 - 40 mg | AZD9567 - 80 mg | AZD9567 - 100 mg | AZD9567 - 125 mg | AZD9567 - 155 mg | Prednisolone - 60 mg | Pooled Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 18 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Cohort 1-8 AZD9567 | 44 (10) | 35 (14) | 35 (8) | 35 (9) | 38 (12) | 34 (9) | 41 (8) | 32 (8) | 0 (0) | 0 (0) | 37 (10)
  Cohort 9 Prenisolone | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 36 (9) | 0 (0) | 36 (9)
  Pooled Placebo | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 37 (11) | 37 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 18 | 72

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of AZD9567 by Assessing the Number of Participants With Adverse Events
Description: Safety and tolerability variables included AEs, vital signs (blood pressure and pulse), ECGs (12-lead ECGs, safety ECGs and telemetry), clinical laboratory safety evaluations (haematology, clinical chemistry [including osteocalcin], coagulation, urinalysis [including 24 hour urine cortisol per day {tU-cortisol}]) and physical examinations.
  Note: No clinically relevant findings were noted in clinical laboratory results and vial signs assessments. Hence, none of the laboratory or vital signs findings were reported as AEs.
Time Frame: At screening, Day -2, Day -1, Day 1 (at pre-dose; 3 & 12 hours post-dose), Day 2 (24 hours post-dose), Day 3 and follow-up (7 to 10 days post-dose)
Population: All participants who received at least one dose of IMP and for whom any safety post-dose data were available were included in the safety analysis for the study. IMP includes AZD9567, Prednisolone 60 mg and placebo.
Measure: Number; unit: Participants
Arm/Group | AZD9567 - 2 mg | AZD9567 - 10 mg | AZD9567 - 20 mg | AZD9567 - 40 mg | AZD9567 - 80 mg | AZD9567 - 100 mg | AZD9567 - 125 mg | AZD9567 - 155 mg | Prednisolone - 60 mg | Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 18
Participants
  Any AE | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 3
  Any AE (including events with outcome =death) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any serious adverse event (SAE) (including death) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any AE leading to discontinuation of AZD9567 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Rate and Extent of Absorption of Single Ascending Doses of AZD9567 by Assessment of Observed Maximum Plasma Concentration (Cmax)
Description: To assess the Cmax of AZD9567 oral suspension following 8 single ascending doses (2, 10, 20, 40, 80, 100, 125 and 155 mg) in Cohorts 1 to 8 in the fasted state. Cmax was taken directly from the individual concentration-time curve.
Time Frame: On Day 1 (at pre-dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12 and 16 hours post-dose), Day 2 (24 hours post-dose) and Day 3 (48 hours post-dose)
Population: The pharmacokinetic (PK) analysis set consisted of all participants in the safety analysis set who received a dose of AZD9567 and had at least one of the parameters Cmax, AUC / AUC(0-last) evaluable. All protocol deviations were considered for the severity/impact and were accounted when participants were assigned to the PK analysis sets.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | AZD9567 - 2 mg | AZD9567 - 10 mg | AZD9567 - 20 mg | AZD9567 - 40 mg | AZD9567 - 80 mg | AZD9567 - 100 mg | AZD9567 - 125 mg | AZD9567 - 155 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nmol/L | 184.9 (20.18) | 751.6 (25.03) | 1327 (17.28) | 2536 (38.33) | 4261 (13.88) | 5835 (14.14) | 6080 (21.30) | 6900 (33.97)
Statistical Analysis 1: Comparison: AZD9567 - 2 mg vs AZD9567 - 10 mg vs AZD9567 - 20 mg vs AZD9567 - 40 mg vs AZD9567 - 80 mg vs AZD9567 - 100 mg vs AZD9567 - 125 mg vs AZD9567 - 155 mg; Test type: Superiority or Other; Slope = 0.847, 90% CI 2-sided [0.807 to 0.887], Standard Error of Mean 0.0238

3. Primary Outcome: Rate and Extent of Absorption of Single Ascending Doses of AZD9567 by Assessment of Time to Reach Maximum Plasma Concentration(Tmax)
Description: To assess the tmax of AZD9567 oral suspension following 8 single ascending doses (2, 10, 20, 40, 80, 100, 125 and 155 mg) in Cohorts 1 to 8 in the fasted state. tmax was taken directly from the individual concentration-time curve.
Time Frame: as for outcome 2
Population: The PK analysis set consisted of all participants in the safety analysis set who received a dose of AZD9567 and had at least one of the parameters Cmax, AUC / AUC(0-last) evaluable. All protocol deviations were considered for the severity/impact and were accounted when participants were assigned to the PK analysis sets.
Measure: Median (Full Range); unit: Hours
Arm/Group | AZD9567 - 2 mg | AZD9567 - 10 mg | AZD9567 - 20 mg | AZD9567 - 40 mg | AZD9567 - 80 mg | AZD9567 - 100 mg | AZD9567 - 125 mg | AZD9567 - 155 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours | 0.50 (20.18) [0.48 to 0.50] | 0.75 (25.03) [0.27 to 1.00] | 0.51 (17.28) [0.50 to 1.50] | 0.75 (38.33) [0.50 to 1.00] | 1.00 (13.88) [1.00 to 1.50] | 1.00 (14.14) [0.50 to 1.50] | 1.00 (21.30) [0.50 to 1.50] | 1.25 (33.97) [0.58 to 2.00]

4. Primary Outcome: Rate and Extent of Absorption of Single Ascending Doses of AZD9567 by Assessment of Terminal Half-life (t½λz)
Description: To assess t½λz of AZD9567 oral suspension following 8 single ascending doses (2, 10, 20, 40, 80, 100, 125 and 155 mg) in Cohorts 1 to 8 in the fasted state. t½λz was estimated as (ln2)/λz.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | AZD9567 - 2 mg | AZD9567 - 10 mg | AZD9567 - 20 mg | AZD9567 - 40 mg | AZD9567 - 80 mg | AZD9567 - 100 mg | AZD9567 - 125 mg | AZD9567 - 155 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours | 4.716 (0.8182) [3.46 to 5.89] | 5.444 (2.157) [2.70 to 9.22] | 3.929 (1.237) [3.13 to 6.31] | 4.199 (1.417) [2.28 to 6.13] | 5.286 (1.469) [3.50 to 6.97] | 5.297 (1.041) [3.89 to 7.02] | 4.664 (1.052) [3.49 to 6.16] | 6.449 (1.778) [4.64 to 8.90]

5. Primary Outcome: Rate and Extent of Absorption of Single Ascending Doses of AZD9567 by Assessment of Area Under the Plasma Concentration-curve From Time Zero to the Time of Last Quantifiable Analyte Concentration (AUC(0-last))
Description: To assess AUC(0-last) of AZD9567 oral suspension following 8 single ascending doses (2, 10, 20, 40, 80, 100, 125 and 155 mg) in Cohorts 1 to 8 in the fasted state.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | AZD9567 - 2 mg | AZD9567 - 10 mg | AZD9567 - 20 mg | AZD9567 - 40 mg | AZD9567 - 80 mg | AZD9567 - 100 mg | AZD9567 - 125 mg | AZD9567 - 155 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*nmol/L | 940.6 (40.32) [3.46 to 5.89] | 5069 (41.83) [2.70 to 9.22] | 7598 (28.12) [3.13 to 6.31] | 13860 (62.81) [2.28 to 6.13] | 31600 (34.57) [3.50 to 6.97] | 41850 (27.82) [3.89 to 7.02] | 40930 (14.32) [3.49 to 6.16] | 56940 (36.80) [4.64 to 8.90]
Statistical Analysis 1: Comparison: AZD9567 - 2 mg vs AZD9567 - 10 mg vs AZD9567 - 20 mg vs AZD9567 - 40 mg vs AZD9567 - 80 mg vs AZD9567 - 100 mg vs AZD9567 - 125 mg vs AZD9567 - 155 mg; Test type: Superiority or Other; Slope = 0.930, 90% CI 2-sided [0.869 to 0.991], Standard Error of Mean 0.0364

6. Primary Outcome: Rate and Extent of Absorption of Single Ascending Doses of AZD9567 by Assessment of Area Under the Plasma Concentration-curve From Time Zero Extrapolated to Infinity (AUC)
Description: To assess AUC of AZD9567 oral suspension following 8 single ascending doses (2, 10, 20, 40, 80, 100, 125 and 155 mg) in Cohorts 1 to 8 in the fasted state. AUC was estimated by AUC(0-last) + Clast/λz. Clast - the last observed quantifiable concentration.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | AZD9567 - 2 mg | AZD9567 - 10 mg | AZD9567 - 20 mg | AZD9567 - 40 mg | AZD9567 - 80 mg | AZD9567 - 100 mg | AZD9567 - 125 mg | AZD9567 - 155 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*nmol/L | 1007 (38.22) [3.46 to 5.89] | 5266 (42.57) [2.70 to 9.22] | 7670 (28.26) [3.13 to 6.31] | 14000 (62.53) [2.28 to 6.13] | 31840 (34.55) [3.50 to 6.97] | 42080 (27.83) [3.89 to 7.02] | 41290 (14.63) [3.49 to 6.16] | 57500 (37.51) [4.64 to 8.90]
Statistical Analysis 1: Comparison: AZD9567 - 2 mg vs AZD9567 - 10 mg vs AZD9567 - 20 mg vs AZD9567 - 40 mg vs AZD9567 - 80 mg vs AZD9567 - 100 mg vs AZD9567 - 125 mg vs AZD9567 - 155 mg; Test type: Superiority or Other; Slope = 0.917, 90% CI 2-sided [0.856 to 0.978], Standard Error of Mean 0.0364

7. Secondary Outcome: Secondary Outcome: Relative Change From Baseline of AUC0-4h for Plasma Glucose to Assess the Effects on Glucose Homeostasis (Oral Glucose Tolerance Test [OGTT])
Description: To assess the effect of AZD9567 and prednisolone on OGTT after administration of 75 g glucose solution, blood samples were collected pre glucose intake and at post glucose intake for the analyses of plasma glucose. AUC0-4h relative change between Day 1 and Day -1 was calculated for each subject in a specific treatment group.
  Note: Total AUC0-4h was calculated using the linear trapezoidal method. Statistical analysis for the change in OGTT plasma glucose total AUC0-4h values were assessed via an analysis of variance (ANCOVA), with treatment as fixed effect.
Time Frame: At Day -1 (baseline) and Day 1 (pre glucose intake and at 30, 60, 90, 120, 150, 180 and 240 minutes post glucose intake)
Population: The pharmacodynamics (PD) analysis set consisted of all participants who received a dose of AZD9567/placebo and who had at least one pre-dose and one post-dose measurement for one of plasma glucose, insulin and C-peptide, and who had no major protocol deviations thought to have impacted the analysis of the PD data.
Measure: Geometric Mean (95% Confidence Interval); unit: min*mmol/L
Arm/Group | AZD9567 - 2 mg | AZD9567 - 10 mg | AZD9567 - 20 mg | AZD9567 - 40 mg | AZD9567 - 80 mg | AZD9567 - 100 mg | AZD9567 - 125 mg | AZD9567 - 155 mg | Prednisolone - 60 mg | Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 18
min*mmol/L | 1.04 [0.963 to 1.12] | 1.01 [0.932 to 1.09] | 1.07 [0.990 to 1.15] | 1.06 [0.986 to 1.14] | 1.08 [0.999 to 1.16] | 1.17 [1.09 to 1.26] | 1.16 [1.08 to 1.25] | 1.20 [1.12 to 1.30] | 1.19 [1.11 to 1.29] | 1.01 [0.964 to 1.05]
Statistical Analysis 1: Comparison: AZD9567 - 2 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 1.03, 90% CI 2-sided [0.960 to 1.11]
Statistical Analysis 2: Comparison: AZD9567 - 10 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 1.00, 90% CI 2-sided [0.929 to 1.08]
Statistical Analysis 3: Comparison: AZD9567 - 20 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 1.06, 90% CI 2-sided [0.987 to 1.14]
Statistical Analysis 4: Comparison: AZD9567 - 40 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 1.06, 95% CI 2-sided [0.983 to 1.13]
Statistical Analysis 5: Comparison: AZD9567 - 80 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 1.07, 90% CI 2-sided [0.995 to 1.15]
Statistical Analysis 6: Comparison: AZD9567 - 100 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 1.17, 90% CI 2-sided [1.09 to 1.25]
Statistical Analysis 7: Comparison: AZD9567 - 125 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 1.15, 90% CI 2-sided [1.07 to 1.24]
Statistical Analysis 8: Comparison: AZD9567 - 155 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 1.20, 90% CI 2-sided [1.11 to 1.29]
Statistical Analysis 9: Comparison: Prednisolone - 60 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 1.19, 90% CI 2-sided [1.11 to 1.27]

8. Secondary Outcome: Relative Change From Baseline of AUC0-4h for Serum Insulin to Assess the Effects on Glucose Homeostasis (Oral Glucose Tolerance Test [OGTT])
Description: To assess the effect of AZD9567 and prednisolone on OGTT after administration of 75 g glucose solution, blood samples were collected pre glucose intake and at post glucose intake for the analyses of serum insulin. AUC0-4h relative change between Day 1 and Day -1 was calculated for each subject in a specific treatment group.
  Note: Total AUC0-4h was calculated using the linear trapezoidal method. Statistical analysis for the change in OGTT serum insulin total AUC0-4h values were assessed via an analysis of variance (ANCOVA), with treatment as fixed effect.
Time Frame: as for outcome 7
Population: The PD analysis set consisted of all participants who received a dose of AZD9567/placebo and who had at least one pre-dose and one post-dose measurement for one of plasma glucose, insulin and C-peptide, and who had no major protocol deviations thought to have impacted the analysis of the PD data.
Measure: Geometric Mean (95% Confidence Interval); unit: min*pmol/L
Arm/Group | AZD9567 - 2 mg | AZD9567 - 10 mg | AZD9567 - 20 mg | AZD9567 - 40 mg | AZD9567 - 80 mg | AZD9567 - 100 mg | AZD9567 - 125 mg | AZD9567 - 155 mg | Prednisolone - 60 mg | Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 18
min*pmol/L | 1.19 [0.987 to 1.45] | 1.20 [0.990 to 1.45] | 1.03 [0.838 to 1.28] | 1.04 [0.863 to 1.26] | 0.999 [0.824 to 1.21] | 0.980 [0.811 to 1.18] | 1.15 [0.953 to 1.39] | 1.16 [0.958 to 1.40] | 0.784 [0.648 to 0.947] | 1.14 [1.02 to 1.27]
Statistical Analysis 1: Comparison: AZD9567 - 2 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 1.05, 90% CI 2-sided [0.872 to 1.26]
Statistical Analysis 2: Comparison: AZD9567 - 10 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 1.05, 90% CI 2-sided [0.874 to 1.26]
Statistical Analysis 3: Comparison: AZD9567 - 20 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 0.907, 90% CI 2-sided [0.745 to 1.10]
Statistical Analysis 4: Comparison: AZD9567 - 40 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 0.914, 90% CI 2-sided [0.762 to 1.10]
Statistical Analysis 5: Comparison: AZD9567 - 80 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 0.876, 90% CI 2-sided [0.728 to 1.05]
Statistical Analysis 6: Comparison: AZD9567 - 100 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 0.860, 90% CI 2-sided [0.716 to 1.03]
Statistical Analysis 7: Comparison: AZD9567 - 125 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 1.01, 90% CI 2-sided [0.842 to 1.21]
Statistical Analysis 8: Comparison: AZD9567 - 155 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 1.02, 90% CI 2-sided [0.846 to 1.22]
Statistical Analysis 9: Comparison: Prednisolone - 60 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 0.687, 90% CI 2-sided [0.572 to 0.825]

9. Secondary Outcome: Relative Change From Baseline of AUC0-4h for Serum C-peptide to Assess the Effects on Glucose Homeostasis (Oral Glucose Tolerance Test [OGTT])
Description: To assess the effect of AZD9567 and prednisolone on OGTT after administration of 75 g glucose solution, blood samples were collected pre glucose intake and at post glucose intake for the analyses of serum C-peptide. AUC0-4h relative change between Day 1 and Day -1 was calculated for each subject in a specific treatment group.
  Note: Total AUC0-4h was calculated using the linear trapezoidal method. Statistical analysis for the change in OGTT serum C-peptide total AUC0-4h values were assessed via an analysis of variance (ANCOVA), with treatment as fixed effect.
Time Frame: as for outcome 7
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: min*nmol/L
Arm/Group | AZD9567 - 2 mg | AZD9567 - 10 mg | AZD9567 - 20 mg | AZD9567 - 40 mg | AZD9567 - 80 mg | AZD9567 - 100 mg | AZD9567 - 125 mg | AZD9567 - 155 mg | Prednisolone - 60 mg | Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 18
min*nmol/L | 1.06 [0.929 to 1.22] | 1.04 [0.913 to 1.19] | 1.02 [0.895 to 1.17] | 0.933 [0.816 to 1.07] | 0.919 [0.804 to 1.05] | 1.00 [0.879 to 1.15] | 0.983 [0.861 to 1.12] | 0.968 [0.846 to 1.11] | 0.749 [0.655 to 0.856] | 1.08 [1.00 to 1.17]
Statistical Analysis 1: Comparison: AZD9567 - 2 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 0.982, 90% CI 2-sided [0.861 to 1.12]
Statistical Analysis 2: Comparison: AZD9567 - 10 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 0.961, 90% CI [0.846 to 1.09]
Statistical Analysis 3: Comparison: AZD9567 - 20 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 0.942, 90% CI 2-sided [0.829 to 1.07]
Statistical Analysis 4: Comparison: AZD9567 - 40 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 0.861, 90% CI 2-sided [0.757 to 0.979]
Statistical Analysis 5: Comparison: AZD9567 - 80 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 0.848, 90% CI 2-sided [0.745 to 0.964]
Statistical Analysis 6: Comparison: AZD9567 - 100 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 0.927, 90% CI 2-sided [0.815 to 1.05]
Statistical Analysis 7: Comparison: AZD9567 - 125 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 0.907, 90% CI 2-sided [0.798 to 1.03]
Statistical Analysis 8: Comparison: AZD9567 - 155 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 0.893, 90% CI 2-sided [0.784 to 1.02]
Statistical Analysis 9: Comparison: Prednisolone - 60 mg vs Pooled Placebo; Test type: Superiority or Other; Ratio (Active Vs Placebo) = 0.691, 90% CI [0.608 to 0.785]

ADVERSE EVENTS:
Time Frame: At screening, Day -2, Day -1, Day 1 (at pre-dose; 3 & 12 hours post-dose), Day 2 (24 hours post-dose), Day 3 and follow-up (7 to 10 days after dose)
Description: Standard adverse event collection. An adverse event is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product
Arm/Group | AZD9567 - 2 mg | AZD9567 - 10 mg | AZD9567 - 20 mg | AZD9567 - 40 mg | AZD9567 - 80 mg | AZD9567 - 100 mg | AZD9567 - 125 mg | AZD9567 - 155 mg | Prednisolone - 60 mg | Pooled Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/18
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 1/6 | 0/6 | 0/6 | 2/6 | 1/6 | 0/6 | 0/6 | 3/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD9567 - 2 mg (N=6) | AZD9567 - 10 mg (N=6) | AZD9567 - 20 mg (N=6) | AZD9567 - 40 mg (N=6) | AZD9567 - 80 mg (N=6) | AZD9567 - 100 mg (N=6) | AZD9567 - 125 mg (N=6) | AZD9567 - 155 mg (N=6) | Prednisolone - 60 mg (N=6) | Pooled Placebo (N=18)
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All clinical study findings and documents will be regarded as confidential. The investigator and members of his/her research team must not disclose such information without prior written approval from the sponsor.